CLINICAL TRIAL: NCT05818878
Title: Prospective, Multicentric Study to Assess Stability of a Tapered Porous Coated Stem and a Cementless Hemispherical Acetabular Component
Brief Title: RSA Masterloc Study Australia
Status: Active, not recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.018.01
Record Dates: First submitted 2023-04-05; First posted 2023-04-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Radiostereometric Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective, multicentric study that aim to assess stability of a tapered porous coated stem and a cementless hemispherical acetabular component.

Main Translation and rotation around the x., y-, and z-axis of the femoral and cup component by radiostereometric analysis (RSA) at immediate post op (within 5 days and before weight bearing), 6 months, 1year and 2 years

DETAILED DESCRIPTION:
Aim of this study is to assess stem and cup migration over the time in patient subjected to a total hip arthroplasty. Medical Device Research Australia will perform image analysis services and reporting for model based radiostereometric analysis (RSA) of cementless fixation of the femoral and acetabular cup components. Migration of the components will be measured with model-based RSA (MBRSA) at immediate post op (within 5 days and before weight bearing), 6 months, 1year and 2 years A subgroup of 26 patients will be invited to be evaluated also by additional RSA analysis: the first 13 patients for each investigator who will accept.

The results of this work will establish the mechanical stability of Masterloc femoral component (Medacta International SA) and MPACT acetabular component (Medacta International SA), provide a general estimate of survivorship, and establish clinical safety and efficacy as measured by RSA and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of the hip necessitating primary hip replacement,
* Suitability for straight cementless stem,
* Adult male and female under 70years old,
* Ability to give informed consent,
* Patients who understand the conditions of the study and are willing to participate for the length of the prescribed follow-up.

Exclusion Criteria:

* Post-traumatic deformity in the affected hip,
* Patient suffering by rheumatoid arthritis,
* Patient suffering by congenital or developmental deformity,
* Severe osteoporosis,
* Earlier surgery in the hip to be operated on,
* Perioperative fracture,
* Personal disorders (dementia, alcohol or drug abuse etc) suspected of making completion of the trial uncertain,
* Patients with a history of active infection
* Pregnant women or those seeking to become pregnant

Max Age: 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 26 patients who entirely fulfil the inclusion/exclusion criteria. The patients will be recruited in a period of 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
RSA imaging | 2 years
  All RSA analysis will be performed Computer Aided Design (CAD) based Roentgen Stereophotogrammetry Analysis (RSA).
  The micro-motion results will be calculated and reported as translations and rotations along and about the three anatomic axes. The subsidence of the hip stem is included in the results. The motion of the femoral stem and acetabular cup will be described in relation to the marker beads placed in the proximal femur and acetabular bone during surgery respectively.
  The first CAD based RSA examination (within 5 days and prior to weight bearing) serves as the reference baseline. All subsequent evaluations of micromotion are related to the relative position of the implanted medical device with respect to the bone (bone markers) at the time of the evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dixon, Medicine, Principal Investigator — Southerland Public Hospital
Locations (1):
- Southerland Public Hospital, Sydney, Australia

IPD SHARING:
Plan to Share IPD: No